CLINICAL TRIAL: NCT02581657
Title: Phase 2a Multicenter, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Response of PE0139 Injection in Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: Study to Assess the Safety, Tolerability, PK and PD Response of PE0139 Injection in Adult Subjects With T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PE0139-PT-CL-0002
Record Dates: First submitted 2015-10-09; First posted 2015-10-21 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PE0139 Injection (Experimental): PE0139 Subcutaneous Injection - 6 weekly doses
  Interventions: Drug: PE0139 Injection
- Placebo Injection (Placebo Comparator): Placebo Subcutaneous Injection - 6 weekly doses
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: PE0139 Injection — PE0139 Injection
  Arms: PE0139 Injection
Drug: Placebo Injection — Placebo Injection
  Arms: Placebo Injection

SUMMARY:
This study is a randomized, double-blind (Investigator and study subject), placebo controlled multiple dose sequential ascending dose study that will enroll up to 47 male and female subjects with type 2 diabetes mellitus (T2DM) in up to four cohorts.

DETAILED DESCRIPTION:
This study is a randomized, double-blind (Investigator and study subject), placebo controlled multiple dose sequential ascending dose study that will enroll up to 47 male and female subjects with T2DM in up to four cohorts; (6 active/2 placebo subjects in cohort 1, and up to 9 active/4 placebo in each subsequent cohort).

This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic response of PE0139 in the presence of existing stable non-insulin antidiabetic background therapy. Subjects will return weekly for a total of 6 doses of study drug.

Study remains active, not recruiting as subjects who received active study drug will be followed for secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent and follow all study-related procedures;
* Male subjects and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study drug;
* Body mass index ≥ 18 kg/m2 and ≤ 45 kg/m2;
* Diagnosed with T2DM with HbA1c of ≥ 7.5% and <11.0% and who is currently taking a non-insulin antidiabetic therapy at stable dose(s) for 3 months prior to screening;
* Willing and able to comply with all study procedures including wearing a continuous glucose monitoring device and performance of frequent self-monitored blood glucose profiles according to the protocol;
* Minimum 7-day average daily glucose of 154 mg/dL (based on CGM) at baseline evaluation;
* Willing to refrain from taking acetaminophen (paracetamol) containing products (e.g., Tylenol®) 24 hours prior to the placement of the CGM device and throughout the time period when the CGM device is worn;
* Live and work in an area with reliable Verizon cellular service for transmission of glucose data required for use of the Telcare Glucose Monitoring System.

Exclusion Criteria:

* Clinical diagnosis of Type 1 diabetes;
* Currently taking or have routinely taken, within 6 months prior to screening, a long or short-acting insulin;
* Self-reported significant change in weight defined as either a loss or gain ≥ 10% during the three month period prior to screening or between screening and randomization;
* Known allergy to, or serious adverse effect caused by an approved, or investigational insulin product or any of its components;
* Currently taking any of the following medications: thiazide or furosemide diuretics, beta-blockers, estrogens or other hormonal replacement therapy, or other chronic medications with known adverse effects on glucose tolerance levels unless the subject has been on stable doses of such agents for at least 2 months prior to screening and have no planned changes in concomitant medication usage during the study period;
* Self-reported history of severe hypoglycemia or hypoglycemic unawareness, as judged by the Investigator;
* Self-reported history of acute complications secondary to diabetes within the last 6 months prior to screening or signs or symptoms of clinically significant diabetes related complications prior to screening;
* Malignant disease defined as: Self-reported history of malignant melanoma or breast cancer; Self-reported history of other types of cancer (excludes basal/squamous cell carcinoma or cervical carcinoma if treated and condition not currently active) within the last 5 years prior to screening;
* Unstable cardiovascular disease defined as one or more of the following: Self-reported history of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to screening; Self-reported history of or currently have NYHA Class III-IV heart failure prior to screening; Self-reported history of unstable angina within 3 months prior to screening; Uncontrolled/sustained hypertension; Self-reported history of clinically significant ECG abnormalities or evidence of clinically significant ECG abnormalities;
* Clinically significant renal and/or hepatic dysfunction noted on safety labs;
* Absolute requirement for corticosteroids or have routinely received systemic steroids within 12 months prior to randomization or use of inhaled corticosteroids within 1 month prior to randomization. A single short course treatment of systemic steroids to treat an acute infection will not exclude the subject if taken more than 3 months from screening;
* Pregnant or lactating female subjects;
* Known history of alcohol abuse or use of illicit drugs within 1 year prior to screening, and/or who test positive for alcohol and illicit drugs prior to randomization. Note: A subject will be considered in violation of the study if they test positive prior to any planned dosing and will be discontinued from the study;
* Positive screening for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies at screening;
* Previously received PE0139;
* Participating in any other study and have received any other investigational medication or device within 30 days prior to screening or are taking part in a non-medication study which, in the opinion of the Investigator, would interfere with the outcome of the study;
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent or would confound the secondary objectives of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (as assessed by incidence and severity of adverse events (AEs), hypoglycemia and changes from baseline in vital signs, ECGs and safety laboratory parameters). | AEs and hypoglycemia (Day -60 to 63), Vital signs (Days -60, -10, 0, 7, 14, 21, 28, 35, 42, 49 and 63), safety laboratory parameters (-60, -10, 14, 28, 42, 49 (as needed), and 63) ECGs (-60, -10, 14, 28, 42, 49 (as needed) and 63).
  To evaluate the safety and tolerability (as assessed by incidence and severity of AEs, hypoglycemia and changes from baseline in vital signs, ECGs and safety laboratory parameters) of multiple ascending doses of PE0139 administered as once weekly injection for 6 weeks in adults with T2DM.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile - Area under the curve over the dosing interval (AUC (0-t)) | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Area under the curve concentration-time profile from 0 to Tmax [AUC (0-tmax)] and from Tmax to t [AUC(tmax-t] | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Maximum serum concentration (Cmax) | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Time to Cmax (Tmax) | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Elimination Rate Constant (Lamda z) | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Elimination half-life (t1/2) | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Clearance (CL/F), uncorrected for bioavailability | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacokinetic (PK) profile - Volume of Distribution (Vz/F), uncorrected for bioavailability | PK measured for Dose 1 (pre-dose, 1, 3, 6 hours post-dose, daily for 6 days), Doses 2-5 given on days 7, 14, 21 and 28, respectively, (pre-dose) and Dose 6 (pre-dose, 1, 3 and 6 hours post dose, daily for 10 days and 14 days post-dose).
  Characterize the PK profile of PE0139 following 6 weeks repeat, once-weekly dosing to explore dose response relationship.
Pharmacodynamic (PD) Profile - Change from baseline in fasting plasma glucose | PD response measured as fasting plasma glucose (FPG) (daily by subject up to day 21 and Days -60, between days -10 and -7, 0, 1-7, 14, 21, 28, 35, 36-49 and 63 at CRU)
  Characterize the PD response of various doses of PE0139 and glucose (as assessed by fasting and non-fasting plasma glucose)
Pharmacodynamic (PD) Profile - Change from baseline in average glucose by CGM | PD response measured by continuous glucose monitoring (CGM) (baseline collected ≥7 days pre-dose daily after dose 3 for 4 weeks)
  Characterize the PD response of various doses of PE0139 and glucose (as assessed by CGM)
Fructosamine changes | Measured at pre-dose and 7 days after last dose
  Assess the effect of various doses of PE0139 on change in fructosamine following 6 weeks of repeat, once-weekly dosing.
Required dose adjustment to background therapy | All scheduled and unscheduled visits (Days -60 to 63)
  Assess the incidence for required dose adjustment to background therapy across various doses of PE0139 and compared to placebo.
Reported hypoglycemic events (% of subjects experiencing severe and non-severe hypoglycemic events) | All scheduled and unscheduled visits (Days -60 to 63)
  Describe incidence, severity, and duration of reported hypoglycemic events across various doses of PE0139 and compared to placebo. Reported as % of subjects experiencing a hypoglycemic event (severe (requiring medical assistance or ≤36 mg/dL glucose) or non-severe (not requiring medical assistance and <70mg/dL glucose))
Binding anti-drug antibodies to PE0139 and insulin (as needed). If positive, neutralizing activity will also be assessed. | Collected at Pre-dose, Days 7, 14, 21, 28, 35, 42, 49, 63 and 91.
  Characterize the immunogenicity profile (binding drug antibodies to PE0139 and insulin (as needed) and neutralizing antibodies if noted to be positive) following 6 weeks of repeat, once-weekly dosing.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - National Research Institute, Huntington Park, California
  - Meridien Research, Bradenton, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Rainier Clinical Research, Renton, Washington